CLINICAL TRIAL: NCT04215965
Title: Efficacy and Safety of a Low-citrate-based Anticoagulation With Calcium-free Phosphate-containing Replacement Fluid Compared to Standard Citrate-based Anticoagulation Protocol in Patients Requiring Continuous Renal Replacement Therapy; a Randomized Controlled Trial
Brief Title: Efficacy and Safety of a Citrate-based Anticoagulation With Calcium-free Phosphate-containing Fluid in Renal Replacement Therapy
Acronym: Phosphorus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-52
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Critical Care
Keywords: CRRT; Renal failure; Citrate; Phosphore
MeSH Terms: conditions — Renal Insufficiency | interventions — Dialysis Solutions; Replantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Standard citrate protocol (Experimental): CVVHDF will be performed using Regiocit solution in the predilution mode, Biphozyl in the dialysate and postdilution mode. CRRT will be started at a dose of 35 ml/kg/h.
  Interventions: Drug: Biphozyl (dialysate and replacement)
- Conventionnal citrate protocol (Active Comparator): CVVHDF will be performed using Regiocit solution in the predilution mode, Prismocal B22 (calcium and phosphate free) in the dialysate mode, and Phoxilium in the postdilution mode. CRRT will be started at a dose of 35 ml/kg/h.
  Interventions: Drug: Prismocal B22 (dialysate) + phoxilium (replacement)

INTERVENTIONS:
Drug: Biphozyl (dialysate and replacement) — Replacement solution with phosphate and without calcium in CRRT with citratre-based antigoagulation
  Arms: Experimental Standard citrate protocol
Drug: Prismocal B22 (dialysate) + phoxilium (replacement) — solution with phosphate and calcium in CRRT with citratre-based antigoagulation
  Arms: Conventionnal citrate protocol

SUMMARY:
In the present prospective multicenter RCT we will evaluate the effects on efficacy, acid-base status and serum phosphate levels of a new RCA protocol for Continuous Venovenous Hemodiafiltration (CVVHDF) using an 18 mmol/l citrate solution in combination with a calcium-free phosphate-containing solution, acting as dialysate and replacement fluid. The new protocol will be introduced with the following targets: a) to refine buffers balance of a previously adopted RCA protocol for Continuous Venovenous Hemofiltration (CVVH), based on a 18 mmol/l citrate solution (Regiocit) combined with calcium and phosphate-free dialysate fluid (PrismOcal B22) and a conventional phosphate-containing replacement fluid (Phoxilium) to prevent CRRT-related phosphate depletion

ELIGIBILITY:
Inclusion Criteria:

1. Acute renal failure requiring CRRT
2. Suitability for regional anticoagulation of the CRRT circuit
3. Clinical equipoise regarding the method of circuit anticoagulation
4. Subject is affiliated with a social security system (if required by individual country regulations).
5. Subject meets national regulatory criteria for clinical trial participation.
6. Subject or subject's Legally Authorized Representative (LAR) has signed the study Informed Consent form

Exclusion Criteria:

1. Age less than 18 years
2. Expected stay in ICU less than 24 hours
3. Pregnant or breastfeeding
4. Suspected ischemic hepatitis or liver failure
5. Chronic kidney disease requiring dialysis prior to ICU admission
6. As applicable by French law, subject who is a protected individual such as an incompetent adult or incarcerated person
7. Metformin and acethaminophen intoxication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-02 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Circuit lifetime | First 3 days of continous renal replacempent therapy
  Number of minutes lifespan circuit

SECONDARY OUTCOMES:
Efficacy of the new RCA solution | first 3 days of CRRT
  Mean daily delivered RRT dose during the first 3 days of CRRT in ml/kg/h between two groups
Efficacy of the new RCA solution | first 3 days of CRRT
  Percentage of decreasing urea during CRRT course between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO, Study Director — Assistance Publique Hopitaux De Marseille

IPD SHARING:
Plan to Share IPD: No